CLINICAL TRIAL: NCT04639583
Title: Utilization of Near-Infrared Spectroscopy Technology to Determine Normative Cerebral Regional Oxygen Saturation in a Preterm Population Born at Altitude
Brief Title: Use of NIRS in Preterm Population Born at Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Jessie R. Maxwell, Assistant Professor of Pediatrics and Neurosciences, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-382
Record Dates: First submitted 2020-11-01; First posted 2020-11-20 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Prematurity; Extreme
MeSH Terms: conditions — Premature Birth | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Intervention Model Description: The study will be a prospective observational study, in which any infant consented to participate in the study will have the NIRS applied for the first 96 hours of life.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Observational Arm (Experimental): Any infant consented to participate in the study will have the NIRS applied for the first 96 hours of life. It will be the goal to apply the NIRS sensors in the first 12 hours of life. All infants will have the same treatment if in the study, but clinicians will not be able to see the data obtained so that there is no clinical interpretation during this time.
  Interventions: Device: Near-infrared spectroscopy (NIRS) utilization

INTERVENTIONS:
Device: Near-infrared spectroscopy (NIRS) utilization — The NIRS devise will be applied so that cerebral regional oxygen saturation (cRSO2) can be measured.

SUMMARY:
Near-infrared spectroscopy (NIRS), is a technology that can provide continuous, non-invasive monitoring of oxygenation in tissue. The objective of this study is to obtain the cerebral regional oxygen saturation (cRSO2) in a preterm population that is born at altitude to determine if the range of "normal" values is different than those obtained at sea level.

ELIGIBILITY:
Inclusion Criteria:

* Infant must be <32 weeks' gestational age at time of delivery.
* Consenting mother/guardian of the infant must speak English. Other languages are not being included due to the need of a translator being brought into the unit, which adds risk to the vulnerable population. Additionally, as the time to consent is a narrow window, adding the complexity of getting a translator may delay the ability to get consent and thus make it more difficult to enroll patients.
* Infants that require blood transfusions during the monitoring time may be included.

Exclusion Criteria:

* Any known cardiac anomaly or other anomaly which may impair perfusion and blood flow.
* Infant born after placental abruption or concern for extreme blood loss immediately after birth.
* Unable to consent the mother/guardian due to maternal health issues after delivering (eg requiring intubation or sedation after the delivery).
* Mothers/guardians that are prisoners, as the study team would like to have continuing communication with the mother during the study period as needed.
* Mothers/guardians that are <18 years of age will not be approached for consent.
* Any mother/guardian that is not able to consent due to having a legal representative will not be approached for consent in this study.
* Any infant that is planned to be placed for adoption
* Infant is greater than 24 hours of age at time of consent.

Ages: 0 Hours to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observational Arm
Started | 21 (21)
NIRS Monitoring | 20
Completed | 20 (20)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Observational Arm
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: weeks] | 28.5 [23.3 to 31.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic latino | 10
  white | 6
  American Indian Alaska Native | 3
  other OR unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 20
rcSO2 (cerebral regional oxygen saturation) [Mean (Inter-Quartile Range); unit: % of rcSO2] | 73.5 [62.5 to 84.5]
CRIB-II (Clinical Risk Index for Babies) II Scoring System [Median (Inter-Quartile Range); unit: score] — CRIB II (clinical risk index for babies, version 2) is a scoring system in prediction of mortality in premature babies (https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4525567/). The score range is 0 to 27, with a better prognosis with lower scores attained.
  score | 8.5 [4.75 to 10]
cFTOE (cerebral fractional tissue oxygen extraction) [Median (Inter-Quartile Range); unit: % of cFTOE] | 21.9 [10.5 to 33.3]

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Regional Oxygen Saturation (cRSO2)
Description: Measure cRSO2 for the first 96 hours of life in infants born preterm.
Time Frame: first 96 hours of life
Measure: Mean (Full Range); unit: percent rcSO2
Arm/Group | Observational Arm
Number analyzed (Participants) | 20
percent rcSO2 | 73.4 [15 to 95]

2. Secondary Outcome: Incidence of Major Complications of Prematurity
Description: Additional items recorded to determine if there is any correlation with the cRSO2 values, including death, intraventricular hemorrhage, necrotizing enterocolitis, sepsis, duration of supplemental oxygen required, time to taking full volume feeds via nippling, and hospital length of stay.
Time Frame: From birth until the end of the birth hospitalization, which would be discharge home or death, whichever occurs first. Estimated time is up to 6 months of age.
Population: Infants with complications of prematurity
Measure: Number; unit: number of infant with condition
Groups:
- Secondary Outcomes IVH: Intraventricular hemorrhage
- Secondary Outcome ROP: Infants requiring treatment for ROP
- Secondary Outcome Sepsis: Infants with late onset sepsis
- Secondary Outcome PDA: Infant with patent ductus arterioles requiring treatment
- Secondary Outcome NEC: Infants diagnosed with necrotizing enterocolitis
Arm/Group | Secondary Outcomes IVH | Secondary Outcome ROP | Secondary Outcome Sepsis | Secondary Outcome PDA | Secondary Outcome NEC
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20
number of infant with condition | 9 | 2 | 3 | 3 | 2

ADVERSE EVENTS:
Time Frame: birth until discharge from birth hospitalization (up to 1 year of age)
Arm/Group | Observational Arm
All-Cause Mortality (participants affected / at risk) | 1/21
Serious Adverse Events (participants affected / at risk) | 19/21
Other Adverse Events (participants affected / at risk) | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observational Arm (N=21)
Intraventricular hemorrhage (Nervous system disorders) | 9 — IVH grade I-IV
Retinopathy of Prematurity (Eye disorders) | 2 — ROP requiring treatment
Necrotizing enterocolitis (Gastrointestinal disorders) | 2 — Infants diagnosed with NEC
Late onset sepsis (Immune system disorders) | 3 — Infants diagnosed with late onset sepsis
Patent Ductus Arteriosus (Cardiac disorders) | 3 — Infants with PDA who required treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT04639583/Prot_SAP_002.pdf
  • Informed Consent Form (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT04639583/ICF_000.pdf